CLINICAL TRIAL: NCT02364037
Title: Implementation of Patient-Centered Contraception Provision in Community Settings
Brief Title: Innovative Model of Patient-Centered ConTraception
Acronym: IMPACCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Family Care Health Centers (Unknown); Memphis Health Center (Unknown); A Step Ahead Foundation (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 201402021; PCORI-CD-12-11-4586 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2015-02-09; First posted 2015-02-16 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Contraception; Unintended Pregnancy
Keywords: intrauterine device; subdermal implant; contraceptive counseling
MeSH Terms: interventions — Intrauterine Devices

STUDY DESIGN:
Intervention Model Description: We used a prospective, controlled time-trend study design, a non-randomized design where outcomes are compared before and after a change in the healthcare setting.
Masking Description: Due to the controlled time-trend design and, therefore, the different time periods for enrollment and follow up for each group, we were unable to mask the research and clinical staff who administered surveys to the study group assignment when collecting data regarding the study outcomes.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase 1: Enhanced Care (Other): Women in Phase 1 of the prospective study will receive the CHOICE Project structured contraceptive counseling in addition to usual care by their health care provider. Contraceptive coverage will be by the usual mechanism such as insurance or financial assistance programs.
  Interventions: Behavioral: CHOICE Project Structured Contraceptive Counseling
- Phase 2: Complete CHOICE (Other): Women in Phase 2 of the prospective study (Complete CHOICE) will receive the CHOICE Project structured contraceptive counseling. Immediately prior to the start of Phase 2, health care providers in participating health centers will undergo a contraceptive education session with a focus on evidence-based guideline for LARC provision and same-day insertion. Participating women will receive cost support for IUDs and implants if she chooses either as her contraceptive method and does not have appropriate insurance coverage.
  Interventions: Behavioral: CHOICE Project Structured Contraceptive Counseling; Behavioral: Contraceptive Education Session; Device: Cost Support for IUDs and implants

INTERVENTIONS:
Behavioral: CHOICE Project Structured Contraceptive Counseling — Women in both phases of the study will receive the structured contraceptive counseling developed by the Contraceptive CHOICE Project.
Behavioral: Contraceptive Education Session — Prior to Phase 2, health care providers at the recruitment sites will undergo a contraceptive education session with a focus on evidence-based provision of contraception including LARC (IUDs and implant) and same-day insertion.
  Arms: Phase 2: Complete CHOICE
Device: Cost Support for IUDs and implants — Women in Phase 2 of the study who desire an IUD or implant can receive one through the study at no cost if they do not have insurance coverage. If women have insurance that covers the device, her insurance will be billed for the cost of the device.
  Arms: Phase 2: Complete CHOICE

SUMMARY:
This study is testing models of contraceptive care that were developed as part of the Contraceptive CHOICE Project. CHOICE is a prospective cohort study of 9,256 women designed to: 1) promote the use of long-acting reversible contraceptive (LARC) methods which include interuterine devices (IUD) and subdermal implants; 2) remove financial barriers to contraception; 3) evaluate continuation of and satisfaction with reversible methods; and 4) reduce unintended pregnancies in the St. Louis region. CHOICE demonstrated that interventions such as comprehensive contraceptive counseling, increased access, and removal of financial barriers increase the uptake of LARC methods and reduce unintended pregnancy. The investigators objective is to determine whether the CHOICE model of contraceptive care can be equally successful in the real world of community clinics.

DETAILED DESCRIPTION:
This project involves comparing two models of contraceptive care; 'enhanced care' which is usual care plus the CHOICE structured contraceptive counseling, and the 'complete CHOICE' group which includes the structured contraceptive counseling as well as provider training and cost support for IUDs and implants. Participants will be enrolled at three partner community clinics by a staff member (site coordinator) dedicated to the research study. All participants will undergo contraceptive counseling as well as a baseline survey with the coordinator. Participants will complete telephone surveys at 3, 6, and 12 months post-enrollment and will be asked about contraceptive method chosen, satisfaction and continuation of the method, and any pregnancies experienced since enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. 14-45 years of age
2. Does not desire pregnancy during the next 12 months
3. Desires reversible contraception
4. Sexually active with a man within the past 6 months or intend to have sex with a man in the next 3 months
5. Willing and able to undergo informed consent
6. Willing to comply with study protocol and 1-year follow-up schedule
7. Not currently pregnant
8. Current patient at Family Care Carondelet, Family Care Forest Park Southeast, Memphis Health Center

Exclusion Criteria:

1. Has undergone a female sterilization procedure such as tubal ligation or hysterectomy
2. Has one sexual partner who has undergone a vasectomy procedure
3. Speaks language other than English or Spanish
4. Currently using an IUD or implant as her contraceptive method

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1008 (Actual)
Dates: Start 2013-08; Primary Completion 2017-01-01 (Actual); Study Completion 2017-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tessa Madden, MD/MPH, Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - Family Care Health Center Forest Park, St Louis, Missouri
  - Family Care Health Center Carondelet, St Louis, Missouri
  - Memphis Health Center, Memphis, Tennessee

REFERENCES:
- [Derived] Madden T, Paul R, Maddipati R, Buckel C, Goodman M, Peipert JF. Comparison of unintended pregnancy at 12 months between two contraceptive care programs; a controlled time-trend design. Contraception. 2019 Sep;100(3):196-201. doi: 10.1016/j.contraception.2019.05.009. Epub 2019 May 24. PMID 31132346
- [Derived] Buckel C, Maddipati R, Goodman M, Peipert JF, Madden T. Effect of staff training and cost support on provision of long-acting reversible contraception in community health centers. Contraception. 2019 Apr;99(4):222-227. doi: 10.1016/j.contraception.2018.12.005. Epub 2019 Jan 24. PMID 30685287

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 2: Complete CHOICE: Women in Phase 2 of the prospective study (Complete CHOICE) will receive the CHOICE Project structured contraceptive counseling. Immediately prior to the start of Phase 2, health care providers in participating health centers will undergo a contraceptive education session with a focus on evidence-based guideline for LARC provision and same-day insertion. Participating women will receive cost support for intrauterine devices (IUDs) and implants if she chooses either as her contraceptive method and does not have appropriate insurance coverage.
Period: Overall Study
Arm/Group | Phase 1: Enhanced Care | Phase 2: Complete CHOICE
Started | 502 | 506
Completed | 458 | 453
Not Completed | 44 | 53
Not completed — Withdrawal by Subject | 7 | 4
Not completed — Lost to Follow-up | 37 | 49

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Enhanced Care | Phase 2: Complete CHOICE | Total
Number analyzed (Participants) | 502 | 506 | 1008
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (6.5) | 26.8 (7.4) | 26.1 (7.0)
Age, Customized [Count of Participants; unit: Participants]
  Age: <20 years old | 88 | 92 | 180
  Age: >=20 years old | 414 | 414 | 828
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 502 | 506 | 1008
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 66 | 105
  Not Hispanic or Latino | 460 | 439 | 899
  Unknown or Not Reported | 3 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 374 | 320 | 694
  Race: White | 96 | 159 | 255
  Race: Other | 32 | 27 | 59
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 502 | 506 | 1008
Education [Count of Participants; unit: Participants]
  =<High School | 317 | 345 | 662
  Some College | 153 | 123 | 276
  =>College Degree | 32 | 38 | 70
Marital Status [Count of Participants; unit: Participants]
  Never Married | 394 | 341 | 735
  Married/Living with Partner | 85 | 132 | 217
  Separated/Divorced/Widowed | 23 | 33 | 56
Federal Poverty Level [Count of Participants; unit: Participants]
  <=100% FPL | 382 | 384 | 766
  101%-200% FPL | 102 | 95 | 197
  >=201% FPL | 16 | 24 | 40
  Unknown or Not Reported | 2 | 3 | 5
Parity [Count of Participants; unit: Participants] — Number of times a participant has given birth
  Participants
    0 | 161 | 165 | 326
    1-2 | 245 | 221 | 466
    3+ | 96 | 120 | 216
Unintended Pregnancy [Count of Participants; unit: Participants]
  At least one prior pregnancy was unintended | 257 | 222 | 479
  No prior pregnancy was unintended | 101 | 147 | 248
  Never pregnant | 143 | 135 | 278
  Missing | 1 | 2 | 3
Insurance Status [Count of Participants; unit: Participants]
  None | 120 | 149 | 269
  Public | 311 | 274 | 585
  Commercial | 70 | 82 | 152
  Missing | 1 | 1 | 2
Participant feelings about becoming pregnant in next 12 months [Count of Participants; unit: Participants]
  Upset | 322 | 293 | 615
  Neutral | 102 | 101 | 203
  Pleased | 49 | 60 | 109
  Unsure | 29 | 52 | 81
Contraceptive method used immediately prior to enrollment visit [Count of Participants; unit: Participants]
  IUD/Implant | 19 | 46 | 65
  Depot Medroxyprogesterone Acetate (DMPA) | 185 | 125 | 310
  Contraceptive Pills/Patch/Ring | 67 | 37 | 104
  Condoms | 46 | 77 | 123
  Other | 19 | 15 | 34
  Nothing | 166 | 206 | 372

OUTCOME MEASURES:

1. Primary Outcome: Unintended Pregnancy
Description: The number of self-reported unintended pregnancies.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Enhanced Care | Phase 2: Complete CHOICE
Number analyzed (Participants) | 502 | 506
Participants | 46 | 25

2. Secondary Outcome: Contraceptive Method Use Upon Enrollment Completion
Description: This measure indicates the contraceptive method that the patient left with after the clinical visit on the day of enrollment. Patients could have received desired new method, received a bridge method, stayed on current method, or received no method.
Time Frame: On the day of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Enhanced Care | Phase 2: Complete CHOICE
Number analyzed (Participants) | 502 | 506
Participants
  Hormonal IUD | 10 | 40
  Copper IUD | 2 | 11
  Implant | 17 | 110
  DMPA | 220 | 145
  Pills/Patch/Ring | 113 | 66
  Condoms | 35 | 57
  Other | 13 | 8
  Nothing | 92 | 69

3. Secondary Outcome: Desired Contraceptive Method at Enrollment Visit
Description: This could be a new method, an existing method, or nothing if participant did not choose a method
Time Frame: On the day of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Enhanced Care | Phase 2: Complete CHOICE
Number analyzed (Participants) | 502 | 506
Participants
  Hormonal IUD | 41 | 85
  Copper IUD | 27 | 26
  Implant | 85 | 162
  DMPA | 192 | 127
  Pills/Patch/Ring | 104 | 53
  Condoms | 13 | 16
  Other | 5 | 2
  Nothing | 35 | 35

4. Secondary Outcome: Participants Choosing Long-Acting Reversible Contraception (LARC) at Enrollment Visit
Description: Number of women choosing an IUD or implant as their preferred contraceptive method
Time Frame: On the day of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Enhanced Care | Phase 2: Complete CHOICE
Number analyzed (Participants) | 502 | 506
Participants | 153 | 273

5. Secondary Outcome: Same Day LARC Insertion
Description: Of the participants who chose LARC as their preferred method, the number who received the device the same day as their enrollment visit.
Time Frame: On the day of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Enhanced Care | Phase 2: Complete CHOICE
Number analyzed (Participants) | 153 | 273
Participants | 21 | 147

ADVERSE EVENTS:
Arm/Group | Phase 1: Enhanced Care | Phase 2: Complete CHOICE
Serious Adverse Events (participants affected / at risk) | 0/502 | 0/506
Other Adverse Events (participants affected / at risk) | 0/502 | 0/506

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No